CLINICAL TRIAL: NCT01376765
Title: Phase I, Double-Blinded, Placebo-Controlled, Dose- Escalation Study of the Safety and Immunogenicity of Recombinant SARS-CoV deltaTM S Protein Vaccine Formulated With and Without Alhydrogel® in Healthy Adults When Administered by the Intramuscular Route
Brief Title: Phase I Dose Escalation SARS-CoV Recombinant S Protein, With and Without Adjuvant, Vaccine Study
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 09-0100
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2012-04

CONDITIONS: SARS
Keywords: SARS, coronavirus, vaccine, adjuvant, Alhydrogel®, severe acute respiratory syndrome
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Coronavirus Infections | interventions — Aluminum Hydroxide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Cohort 1 (Experimental): Recombinant S protein severe acute respiratory syndrome (SARS) vaccine received with aluminum hydroxide adjuvant (Alhydrogel®), without adjuvant, or placebo in 2 intramuscular doses, 28 days apart, at 5 micrograms per dose; 12 subjects receive unadjuvanted vaccine (SARS vaccine alone); 12 subjects receive adjuvanted vaccine {(SARS vaccine with aluminum hydroxide adjuvant (Alhydrogel®)}; 4 subjects receive placebo.
  Interventions: Drug: Aluminum hydroxide adjuvant (Alhydrogel®); Other: Phosphate buffered saline Placebo; Biological: Recombinant S protein SARS vaccine
- Cohort 3 (Experimental): SARS vaccine with adjuvant, without adjuvant, or placebo; l in 2 intramuscular doses, 28 days apart, at 45 micrograms per dose; 12 subjects receive unadjuvanted vaccine (SARS vaccine alone); 12 subjects receive adjuvanted vaccine (SARS vaccine with adjuvant); 4 subjects receive placebo.
  Interventions: Drug: Aluminum hydroxide adjuvant (Alhydrogel®); Other: Phosphate buffered saline Placebo; Biological: Recombinant S protein SARS vaccine
- Cohort 2 (Experimental): SARS vaccine with adjuvant, without adjuvant, or placebo in 2 intramuscular doses, 28 days apart, at 15 micrograms per dose; 12 subjects receive unadjuvanted vaccine (SARS vaccine alone); 12 subjects receive adjuvanted vaccine (SARS vaccine with adjuvant) 4 subjects receive placebo.
  Interventions: Drug: Aluminum hydroxide adjuvant (Alhydrogel®); Other: Phosphate buffered saline Placebo; Biological: Recombinant S protein SARS vaccine

INTERVENTIONS:
Drug: Aluminum hydroxide adjuvant (Alhydrogel®) — Aluminum hydroxide adjuvant (Alhydrogel®);given with SARS vaccine; 2 intramuscular doses, 28 days apart, Cohort 1: 12 subjects given vaccine with adjuvant at 5 micrograms per dose; Cohort 2: 12 subjects given vaccine with adjuvant at 15 micrograms per dose; Cohort 3: 12 subjects given vaccine with adjuvant at 45 micrograms per dose
Other: Phosphate buffered saline Placebo — Phosphate buffered saline Placebo; 2 intramuscular doses, 28 days apart. Cohort 1: 4 subjects given placebo at 5 micrograms per dose; Cohort 2: 4 subjects given placebo at 15 micrograms per dose; Cohort 3: 4 subjects given placebo at 45 micrograms per dose
Biological: Recombinant S protein SARS vaccine — Recombinant S protein severe acute respiratory syndrome (SARS) vaccine given with adjuvant or without adjuvant; 2 intramuscular doses, 28 days apart, Cohort 1: 12 subjects given vaccine only or vaccine with adjuvant at 5 micrograms per dose; Cohort 2: 12 subjects given vaccine only or vaccine with adjuvant at 15 micrograms per dose; Cohort 3: 12 subjects given vaccine only or vaccine with adjuvant at 45 micrograms per dose

SUMMARY:
This is a multi-center, randomized, double-blinded, placebo-controlled, outpatient study. Recombinant deltaTM S Protein Severe Acute Respiratory Syndrome (SARS) Vaccine With and Without Aluminum Hydroxide Adjuvant (Provided through contract N01-AI-30023, manufactured by Protein Sciences Corporation), two doses, administered at 28 day interval. 1. S Protein Severe Acute Respiratory Syndrome (SARS) Vaccine without adjuvant: 5.0, 15.0 and 45.0 mcg per 0.5 ml dose. 2. S Protein SARS Adjuvanted Vaccine: 5.0, 15.0 and 45.0 mcg per 0.5 ml dose. PLACEBO: diluents/placebo without vaccine (Phosphate Buffer Saline (PBS) with lower phosphate concentration). Approximately 84 healthy male and nonpregnant female subjects 18 to 40 years of age will be enrolled.

DETAILED DESCRIPTION:
This is a Phase 1,multi-center, randomized, double-blinded, placebo-controlled, outpatient study in healthy male and nonpregnant female subjects 18 to 40 years of age, inclusive. Three dosing cohorts to investigate the safety, reactogenicity, and immunogenicity of Recombinant S protein Severe Acute Respiratory Syndrome (SARS) vaccine, with and without aluminum hydroxide adjuvant manufactured by Protein Sciences Corporation, administered intramuscularly on Days 0 and 28 at a dose of 5, 15, or 45 mcg; controls will receive the diluents/placebo without vaccine. Approximately 84 subjects are expected to be enrolled. All subjects will receive 2 doses of their assigned treatment via IM injection approximately 28 days apart, followed by assessments at 6, 12, 15, 18, 21 and 24 months after the second dose.

ELIGIBILITY:
Inclusion Criteria:

* Males or nonpregnant females between the ages of 18 and 40 years, inclusive.
* Women of childbearing potential (not surgically sterile via tubal ligation, bilateral oophorectomy or hysterectomy or who have not been postmenopausal for >/=1 year) must agree to practice adequate contraception for the 30-day period before vaccination through 90 days after the second vaccination. Acceptable birth control methods for the purposes of this study may include, but are not limited to, abstinence, monogamous relationship with vasectomized partner, barrier methods such as condoms, diaphragms, spermicides, and intrauterine devices, and licensed hormonal methods.
* In good health, as judged by the investigator and determined by vital signs [temperature < 38 degrees C, heart rate </= 100 bpm and > 50 bpm, systolic blood pressure </= 140 mmHg and > 89 mmHg, diastolic blood pressure </= 90 mmHg and >/= 60 mm Hg, respiratory rate >/= 12 breath per minute and < 17 breaths per minutes (see toxicity table in Section 9.1.2)], medical history and a targeted physical examination, as indicated, based on medical history.
* Screening laboratory values must be within normal limits. These include blood hemoglobin, white blood cell (WBC) count, eosinophils, platelets, absolute eosinophil, neutrophil, and lymphocyte cell counts, creatinine, aspartate aminotransferase (AST), alanine transaminase (ALT), bilirubin (total), glucose (random), and urinalysis (proteinuria and hematuria). See toxicity table in Section 9.1.3.2. Note: creatinine values lower than the normal are acceptable.
* Able to understand and comply with planned study procedures.
* Willing to be available for all study-required procedures, visits and calls for the duration of the study.
* Provide written informed consent before initiation of any study procedures and be available for all study visits.
* Negative for IgG antibodies to S protein of Severe Acute Respiratory Syndrome coronavirus (SARS-CoV) measured by ELISA.
* Negative for antibodies to Human Immunodeficiency Virus (HIV) and hepatitis C virus and for hepatitis B surface antigen.
* Negative for IgG antibodies to S protein of Severe Acute Respiratory Syndrome coronavirus (SARS-CoV) measured by ELISA.
* Negative for antibodies to Human Immunodeficiency Virus (HIV) and hepatitis C virus and for hepatitis B surface antigen.

Exclusion Criteria:

* A known allergy to components of the vaccine.
* A positive serum or urine pregnancy test within 24 hr prior to vaccination (if female of childbearing potential as defined in Inclusion Criterion 2), women who are planning to become pregnant from 30 days prior to entering the study until 90 days after the final study vaccination, or women who are breastfeeding.
* Immunosuppression as result of underlying illness or treatment or use of anticancer chemotherapy or radiation therapy (cytotoxic) within the preceding 36 months.
* An active neoplastic disease (excluding nonmelanoma skin cancer or prostate cancer that is stable in the absence of therapy) or a history of any hematologic malignancy. Nonactive neoplastic disease is defined as no neoplastic disease or treatment for neoplastic disease within the past 5 years.
* A history of autoimmune disease (systemic lupus, rheumatoid arthritis, scleroderma, polyarteritis, thyroiditis, etc).
* Used an immunosuppressive or immunomodulatory drug such as >0.5 mg/kg/day or >/=20 mg total dose/day of prednisone orally or >800 mcg of inhaled beclomethasone for 2 or more consecutive weeks within 6 months prior to the 1st vaccination. (Nasal and topical steroids are allowed.)
* A known human immunodeficiency virus (HIV) infection, or active hepatitis B, or hepatitis C virus infection.
* A diagnosis of schizophrenia, bipolar disease, or other major psychiatric diagnosis in the past 3 years.
* Hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others in the past 3 years.
* Receiving psychiatric drugs listed below*. Subjects who are receiving a single antidepressant drug and are stable for at least 3 months prior to enrollment, without decompensating symptoms will be allowed to be enrolled in the study.

  *aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, trifluopromazine, chlorprothixene, chlorpromazine, perphenazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate, or lithium citrate.
* A history of receiving immunoglobulin or other blood product within the previous 3 months before vaccination.
* Received or plan to receive any live licensed vaccines within 4 weeks or inactivated licensed vaccines within 2 weeks of each vaccination,
* An acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses or is not generally seen in healthy, normal subjects. (This includes, but is not limited to, known cardiac disease, pulmonary disease, liver disease, renal disease, unstable or progressive neurological disorders, diabetes mellitus, and transplant recipients.)
* A history of severe reactions following immunization with vaccines.
* Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month before vaccination in this study or expect to receive an experimental agent during the 24-month study period.
* Any condition that would, in the opinion of the investigator, place them at an unacceptable risk of injury, render them unable to meet the requirements of the protocol, or that may interfere with successful completion of the study.
* A history of alcohol or drug abuse during the previous 1 year; for example, daily excessive alcohol use or frequent binge drinking as determined by the investigator, or chronic marijuana abuse or any other illicit drug use.
* Plans to travel outside North America in the time between the 1st vaccination and 56 days following the first vaccination or have plans to travel to Southeast Asia during their entire study participation.
* Body temperature >/=100.4 F (>/=38.0 C) or acute illness within 3 days before vaccination (subject may be rescheduled).
* Planned or have had a known exposure to the Himalayan palm civet, raccoon dog of Southeast Asia, or Chinese horseshoe bat, including bats that have been shipped from Southeast Asia or that were previously housed with Southeast Asian counterparts.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited local and systemic adverse events (AE)within 8 days after vaccination (Days 0-7 and Days 28-35) | 8 days after vaccination (Days 0-7 and Days 28-35)
Incidence of vaccine-related serious adverse events (SAEs) throughout the duration of the study. | Day 0 to Day 758
Occurrence of laboratory abnormalities at 8 days after vaccination (Days 8 and 36) | 8 days after vaccination (Days 8 and 36)

SECONDARY OUTCOMES:
Immunogenicity: Proportion of subjects achieving a detectable serum neutralizing antibody titer against SARS-CoV in each immunized group 28 days after receipt of the second dose of vaccine (approximately Day 56) | 28 days after receipt of the second dose of vaccine (approximately Day 56)
Immunogenicity: GMT of neutralizing antibody titers against SARS-CoV in each immunized group 28 days after receipt of the second dose of vaccine (Day 56). Measurement will include the Day 56 GMT and the mean fold change (GMT ratio Day 56:Day 0) | 28 days after receipt of the second dose of vaccine (Day 56)
Comparison of rates of unsolicited AEs related to vaccine for all subjects between treatment groups and in the combined cohorts receiving vaccine with aluminum hydroxide adjuvant compared with those receiving vaccine with no adjuvant. | intervals from Days 0-7, Days 0-28, Days 8-28, Days 0-56, Days 29-36, and Days 29-56.
Immunogenicity: Geometric Mean Titer (GMT) of antibody titers (IgG ELISA for S protein of SARS-CoV) 28 days after receipt of the second dose of vaccine (Day 56) at each vaccine dose level, with and without adjuvant | 28 days after receipt of the second dose of vaccine (Day 56)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Iowa - Infectious Disease Clinic, Iowa City, Iowa
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio